CLINICAL TRIAL: NCT06662955
Title: Terminal Knee Extension Exercise Synchronize With Audible Cues on Motor Unit Behavior of Vastus Medialis Muscle in Athletes With Anterior Cruciate Ligament Reconstruction
Brief Title: Exercise With Audible Cues on Motor Unit Behavior in Athletes With Anterior Cruciate Ligament Reconstruction
Acronym: ACLR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Komsak Sinsurin, Asst.Prof.Dr., Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MU-CIRB 2024/242.3009
Record Dates: First submitted 2024-10-25; First posted 2024-10-29 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Therapeutic Exercise; Physical Therapy Techniques; Neuromuscular Function
Keywords: ACLR
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Masking Description: Paticipants are blinded groups allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise without audible cues (Active Comparator): Terminal knee extension exercise without audible cues
  Interventions: Behavioral: Exercise
- Exercise with audible cues (Experimental): Terminal knee extension exercise with audible cues
  Interventions: Behavioral: audible cues

INTERVENTIONS:
Behavioral: audible cues — Terminal knee extension exercise with audible cues
  Other Names: Exercise with audible cues
  Arms: Exercise with audible cues
Behavioral: Exercise — Terminal knee extension exercise
  Arms: Exercise without audible cues

SUMMARY:
The closed kinetic chain (CKC) of terminal knee extension exercise (TKE) is designed to activate VM activity for knee injury training. This CKC exercise is effective for highest recruiting muscle activity, especially safe for post-operative knee surgery. The study of ACL reconstruction rehabilitation guideline suggests that exercises can be applied within the early phase of rehabilitation to prevent knee laxity and less knee pain compared to open chain exercise. Therefore, it is interesting to investigate the effects of TKE exercise synchronized with metronome pace on change of VM motor unit behavior in post operative ACL reconstruction. This study focuses on the immediate effect of 1-seesion TKE and expects that adding metronome during TKE will enhance neuromuscular control of VM and may change motor unit behavior.

DETAILED DESCRIPTION:
This study investigates the effect of exercise with sensory integration technique on neuromuscular control in athletes with anterior cruciate ligament reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants who receive primary ACL reconstruction within 2 weeks with or without meniscus repair
* No or mild resting pain (Numeric rating scale ≤ 3)
* Reconstruction procedures using autograft including hamstrings or bone-patella bone grafts
* Age range 18-35 years (33).
* BMI of 18.5-25 kg/m² (34).
* Tegner activity scale ≥ level 4

Exclusion Criteria:

* Non-weight bearing within 2 weeks after the operation (prescription from surgeon)
* Hearing problem, such as being unable to hear the metronome sound or being unable to synchronize exercises with the metronome correctly
* Limitations in knee extension range caused by joint stiffness evaluated by using passive knee range of motion
* Unable to perform active and passive ≥ 30º knee flexion on the operative side
* History of serious injury or operation of lower back and lower extremities such as fracture
* Lower back or lower extremities pain within 6 months before the study
* On the pain killer medication

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-20 (Actual); Primary Completion 2026-10-19 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Average motor unit firing rate (pulse per second, pps) | From enrollment to the end of treatment at 2 weeks
  Motor unit behavior of vastus medialis muscle: Average motor unit firing rate (pulse per second, pps)

SECONDARY OUTCOMES:
Peak motor unit action potential (mV) | From enrollment to the end of treatment at 2 weeks
  Motor unit behavior of vastus medialis muscle: Peak motor unit action potential (mV)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Mahidol University, Salaya, Changwat Nakhon Pathom, Thailand

IPD SHARING:
Plan to Share IPD: Undecided